CLINICAL TRIAL: NCT06279884
Title: A Multicenter Prospective Clinical Cohort Study on the Pathogen Spectrum of Liver Transplant Recipients Complicated With Infection
Brief Title: A Cohort Study on the Pathogen Spectrum of Liver Transplant Recipients Complicated With Infection
Status: Not yet recruiting | Type: Observational
Sponsor: Zhejiang University (Other)
Collaborators: Beijing Ditan Hospital (Other); Beijing YouAn Hospital (Other); Huashan Hospital (Other); Qilu Hospital of Shandong University (Other)
Responsible Party: Principal Investigator, Jiajia Chen, Chief Physician of the First Affiliated Hospital,Zhejiang University School of Medicine, Zhejiang University
Other Study IDs: 2023YFC2308802-03
Record Dates: First submitted 2024-02-19; First posted 2024-02-28 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-03

CONDITIONS: Liver Transplantation; Transplant Recipients
Keywords: Liver Transplant Recipients; Infection; Pathogen spectrum; Cohort study
MeSH Terms: conditions — Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — According to the characteristics of infection, take blood or body fluids from the corresponding infected site.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to map the pathogen profile of secondary infections in liver transplant recipients, to correlate the basic immune status with the characteristics of the secondary infection pathogen profile, and to establish an early warning system for monitoring secondary infections, so as to explore safe and effective therapeutic modalities to further reduce the morbidity and mortality of liver failure. The main questions it aims to answer are:

* Characterize the distribution of pathogenic bacteria infecting liver transplant recipients.
* Establish a monitoring and early warning system for secondary infections.

DETAILED DESCRIPTION:
Liver transplantation is recognized as the most effective treatment for end-stage liver disease, and China's liver transplantation technology has reached the international level, with survival rates of 90%, 80%, and 70% at 1, 5, and 10 years after surgery, respectively. During the perioperative period of liver transplantation, transplant recipients with preoperative organ dysfunction, high surgical trauma, postoperative application of immunosuppressive drugs, and low anti-infective capacity are highly susceptible to associated infections, which are more likely to occur than in other transplant recipients, and have become an important factor affecting the prognosis of liver transplantation. Foreign studies reported that 18% of postoperative liver transplantation deaths were caused by infections, of which bacterial infections were the most common, followed by viral and fungal infections. In the first month after liver transplantation, the incidence of infection is the highest, and bacterial pneumonia is the most common infection, with a high case fatality rate, and the hospitalization time of the patient is significantly prolonged, and the economic expenditure is increased. Early clarification of the type and distribution of pathogenic bacteria infecting liver transplant recipients and prompt initiation of appropriate anti-infective therapy are essential to improve the survival of liver transplant recipients.

ELIGIBILITY:
Inclusion Criteria:

1. Agree to participate in this study and sign the informed consent form;
2. Be of any gender and aged 18-70 years old;
3. No life-threatening underlying diseases and complications during the perioperative period.
4. Undergo liver transplantation within 24 hours.

Exclusion Criteria:

1.Patients deemed unsuitable by the investigator to participate in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Liver transplant recipients
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Secondary Infections in liver transplant recipients at 4 weeks | 4 weeks
  Site of infection, pathogen results such as blood or body fluid pathogen cultures or Next-generation sequencing(NGS) results.
quick SEPSIS RELATED ORGAN FAILURE ASSESSMENT(qSOFA) at 4 weeks | 4 weeks
  qSOFA consists of 3 items: altered state of consciousness, systolic blood pressure ≤ 100 mmHg, and respiratory rate ≥ 22 respirations/min. 2 or more items, i.e., a qSOFA score of ≥ 2, are considered to be suspicious for sepsis.Higher qSOFA scores are associated with a higher risk of patient death.

SECONDARY OUTCOMES:
Occurrence of secondary infections in liver transplant recipients at 8 weeks, including site of infection, pathogen of infection | 8 weeks
  Site of infection, pathogen results such as blood or body fluid pathogen cultures or Next-generation sequencing(NGS) results.
Occurrence of secondary infections in liver transplant recipients at 12 weeks, including site of infection, pathogen of infection | 12 weeks
  Site of infection, pathogen results such as blood or body fluid pathogen cultures or Next-generation sequencing(NGS) results.
qSOFA score at 8 weeks | 8 weeks
  qSOFA consists of 3 items: altered state of consciousness, systolic blood pressure ≤ 100 mmHg, and respiratory rate ≥ 22 respirations/min. 2 or more items, i.e., a qSOFA score of ≥ 2, are considered to be suspicious for sepsis.Higher qSOFA scores are associated with a higher risk of patient death.
qSOFA score at 12 weeks | 12 weeks
  qSOFA consists of 3 items: altered state of consciousness, systolic blood pressure ≤ 100 mmHg, and respiratory rate ≥ 22 respirations/min. 2 or more items, i.e., a qSOFA score of ≥ 2, are considered to be suspicious for sepsis.Higher qSOFA scores are associated with a higher risk of patient death.

CONTACTS AND LOCATIONS:
Overall Officials: Jiajia Chen, Principal Investigator — Zhejiang University